CLINICAL TRIAL: NCT05794022
Title: CoHort of Patients to Identify Biological and Imaging markerS of CardiovascUlar Outcomes in ST Elevation Myocardial Infarction
Brief Title: Cohort of STEMI Patients 2
Acronym: HIBISCUS STEMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL22_0991
Record Dates: First submitted 2023-02-06; First posted 2023-03-31 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; bio-collection; Imaging markers; biomarkers; STEMI; clinical outcomes
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort group (Other): patient with ST-segment elevation myocardial infarction.
  Interventions: Other: MRI; Biological: Biocollection; Behavioral: Quality of life questionaries

INTERVENTIONS:
Other: MRI — 1 MRI at 1 month with gadolinium injection
Biological: Biocollection — Biocollection from blood (H0, H4, H24, H48, 1 month, 1 year), urine (H48) and faecal (initial hospitalisation) samples.
Behavioral: Quality of life questionaries — EQ-5D-5L and HAD questionaries at 1 month and 1 year.

SUMMARY:
ST-segment elevation myocardial infarction (STEMI) is an acute condition that accounts for 75% of sudden deaths in adults over 35 years of age and more than half of all cases of chronic heart failure. However, the mechanism of myocardial infarction remains poorly understood. At present, there is no national information system for myocardial infarction, as there is for other diseases such as multiple sclerosis (OFSEP cohort).

The purpose of this cohort is to enable studies and research projects to be carried out on the descriptive epidemiology of myocardial infarction, monitoring of patients undergoing treatment (safety, efficacy), quality of life and functional consequences of infarction, and research into new biological and imaging prognostic biomarkers. Its general objective is to provide researchers, hospital practitioners, medical interns, academics or industrialists with a quality epidemiological tool for research.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of STEMI defined by ST segment elevation ≥ 0.2 mV in 2 contiguous leads on a 12-lead ECG.
* Management in primary ACT
* Prior oral informed consent followed by signed informed consent as soon as possible.

Exclusion Criteria:

* Diagnosis of STEMI not confirmed on angiography
* Inability to give the subject informed information
* Lack of coverage by a social security scheme
* Obvious contraindication to injected magnetic resonance imaging (claustrophobia, pacemaker, defibrillator, or a metallic body (ferromagnetic), severe renal insufficiency (GFR<30 ml/min), known allergy to the contrast medium ....)
* Pregnant woman or woman of childbearing age without effective contraception, breastfeeding woman.
* Deprivation of civil rights (curators, guardianship, safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2031-06-03 (Estimated); Study Completion 2031-06-03 (Estimated)

PRIMARY OUTCOMES:
Research of potential new markers | 1 year
  Biomarkers assays (prognosis and diagnosis) between inclusion and one-year follow-up (H0, H4, H24, H48, M1, M12 since emergency revascularisation)

SECONDARY OUTCOMES:
Calculation of infarct size on MRI | 1 month
  Measurement of reperfusion lesions on MRI (mass in grams)
Pharmacoepidemiology of myocardial infarction. | 5 years
  Description and evolution of patients' medical treatment between hospital discharge and 5 years follow-up.
Events between inclusion and 5 years follow-up | 5 years
  Time to a major adverse cardiovascular event

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hospices Civils de Lyon - Hôpital Louis Pradel, Bron, Rhone
  - Hospices Civils de Lyon - Hôpital de la Croix Rousse, Lyon, Rhone

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stevic N, Pinede A, Mewton N, Ovize M, Argaud L, Lecour S, Boiteux C, Bochaton T, Cour M. Effect of ventricular fibrillation on infarct size after myocardial infarction: a translational study. Basic Res Cardiol. 2024 Dec;119(6):911-921. doi: 10.1007/s00395-024-01091-9. Epub 2024 Nov 23. PMID 39579225